CLINICAL TRIAL: NCT05860582
Title: A Study of [14C]GB491 on Mass Balance and Biotransformation in Chinese Male Healthy Subjects
Brief Title: A Study of [14C]GB491 in Male Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GB491-MB
Record Dates: First submitted 2023-04-23; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]GB491 (Experimental)
  Interventions: Drug: [14C]GB491

INTERVENTIONS:
Drug: [14C]GB491 — A single 150mg dose of GB491 containing approximately 50 uCi of [14C]GB491.

SUMMARY:
This is an open-label, single-center study to evaluate the mass-balance and pharmacokinetics of GB491 in 4-8 healthy male subjects receiving a single oral 150mg dose of GB491 containing approximately 50 uCi of [14C]GB491. This study will help understand how the drug appears in the blood, urine, and feces after it is administered.

In addition, this study will also evaluate the safety of a single dose of [14C]GB491 when given to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male volunteer between 18 and 50 years of age inclusive
* A total body weight >=50kg, and a BMI of 19.0-26.0 kg/m2
* A signed informed consent document

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease
* Subjects with HBsAg-positive, or HCV-Ab-positive, or TPPA-positive, or HIV infection
* Subjects with a history of habitual constipation/diarrhea, irritable bowel syndrome, or inflammatory bowel disease

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Total radioactivity in plasma PK | Up to 168 hours post dose
  To investigate the distribution ratio of total radioactivity in whole blood to plasma and pharmacokinetic characteristics of total radioactivity in plasma in healthy subjects after a single dose of [14C]GB491.
Total radioactivity in urine and fecal samples | Up to 360 hours post dose
  Quantitative analysis of total radioactivity in urine or feces in healthy subjects after a single dose of [14C]GB491.
Metabolite G1T30 and other major matabolites (if applicable) | Up to 168 hours post dose
  Identify the main metabolites in healthy subjects after oral administration of [14C]GB491 to determine the main biotransformation pathway

SECONDARY OUTCOMES:
Quantitative analysis of drug concentrations of GB491, metabolite G1T30 and other major metabolites (if applicable) in plasma | Up to 168 hours post dose
Adverse events | Up to 360 hours post dose
  The safety of healthy subjects after a single dose of [14C]GB491

CONTACTS AND LOCATIONS:
Overall Officials: Fang HOU, Master, Principal Investigator — Beijing GoBroad Boren Hospital
Locations (1):
- Beijing GoBroad Boren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No